CLINICAL TRIAL: NCT03803878
Title: Medical, Epidemiologic, and Social Aspects of Aging (MESA) Urinary Incontinence Questionnaire: Translation and Validation of the Chinese Language Version in Women With Urgency-predominant Mixed Urinary Incontinence
Brief Title: Translation and Validation of MESA Questionnaire of Chinese Language Version
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principle investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 2018-162-KY
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Questionnaire; Mixed Urinary Incontinence; Urgency-predominant Mixed Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 is anticipated to consist of 300 women with MUI, and the categorization function of MESA questionnaire will be validated among those patients.
- Group 2: Group 2 is anticipated to consist of 282 women with urgency-predominant MUI.
- Group 3: Group 3 is anticipated to consist of 94 women with urgency-predominant MUI.

SUMMARY:
The study is to translate the Medical, Epidemiologic, and Social aspects of Aging (MESA) urinary incontinence questionnaire into a Chinese language version and test the reliability and validity among women with urgency-predominant mixed urinary incontinence.

The hypothesis is that the Chinese language version of the MESA questionnaire will have adequate measurement properties (e.g. reliability and validity).

DETAILED DESCRIPTION:
Mixed urinary incontinence(MUI) is regarded as urgency-predominant when urgency incontinence episodes dominate over stress incontinence episodes, and vice versa. The treatment of MUI often begins with the most bothersome symptoms.

MESA questionnaire is a reliable and validated tool to evaluate the severity and predominance of stress or urgency urinary incontinence. At present, it hasn't been translated into a Chinese language version and validated.

The validation study of MESA questionnaire is embedded in a randomized controlled trial conducted among female patients, of which the data will be collected and analysed.

ELIGIBILITY:
Inclusion criteria

1. Female patients diagnosed with MUI in accordance with EAU guideline by history taking, physical examination, laboratory tests and specialist diagnosis;
2. Age between 18 and 80 years old;
3. At least 4 episodes of UUI in 3-day voiding diary;
4. With MUI for at least 3 months, and urgency urinary incontinence dominates more than 50% of the total incontinence episodes in 3-day voiding diary;
5. Positive cough test;
6. A voluntarily-signed written informed content. For patients in group 1, inclusion criteria of 1), 2), 5) and 6) are required to meet. Those also meeting the criteria of 3) and 4) will enter group 2 at the same time.

For patients in group 2 and groups 3, all inclusion criteria are required to meet.

Exclusion criteria

1. Having pure SUI, pure UUI, overflow UI or neurogenic bladder;
2. Uncontrolled urinary tract infection;
3. Tumor in urinary system or pelvic organs;
4. Pelvic organ prolapse≥degreeⅡ;
5. Residual urine volume≥100ml;
6. Maximum flow rate<15ml/s;
7. In the past 1 month, receiving treatment of acupuncture or positive medications targeted at incontinence, such as antimuscarinic drugs;
8. Underwent anti-incontinence or pelvic organ surgery, including metrectomy;
9. Complication of severe diabetes or hypertension;
10. Complication of diseases in nervous system that could hamper hypourethral function, such as multiple sclerosis, senile dementia, Parkinson's disease, spinal cord injury, cauda equina nerve injury and multiple system atrophy;
11. Severe complications in cardiac, lungs, cerebrum, hepar, renal system, psychonosology and coagulation function, or obvious cognitive disability;
12. Installed a cardiac pacemaker;
13. Allergic to Solifenacin or with contraindications to antimuscarinic drug, including urinary retention, gastrointestinal peristalsis paralysis, myasthenia gravis, ulcerative colitis and angle-closure glaucoma;
14. Allergic to metal or intolerant to the stimulation of electroacupuncture;
15. Pregnant or plan to conceive in the future 1 year, or delivery in the past one year.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The questionnaire validation is targeted at women with urgency-predominant mixed urinary incontinence.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The criteria validity of MESA questionnaire compared with extended clinical evaluation in deciding predominant components of MUI. | screening and baseline periods
  The extended clinical evaluation mainly includes physical examination, 3-day voiding diary, cough stress teat, urinalysis and residual urine volume by ultrasonography.

SECONDARY OUTCOMES:
The criteria validity of MESA questionnaire compared with International Consultation on Incontinence Questionnaire Short Form (ICIQ SF) in severity assessing among women with urgency-predominant mixed urinary incontinence. | baseline
  ICIQ SF is a validated questionnaire to evaluate both the severity of incontinence symptoms and influence on QoL in the past four weeks. The questionnaire is consisted of four items, including frequency, leakage amount, impact on QoL and the cause of urinary incontinence. The total score of the ICIQ SF ranges from 0 to 21, with a higher score indicating worse symptoms and QoL.
The criteria validity of MESA questionnaire compared with 3-day voiding diary in severity assessing among women with urgency-predominant mixed urinary incontinence. | baseline
  In 3-day voiding diary, the type and episodes of incontinence are all recorded.
The test-retest reliability of MESA questionnaire | screening and baseline periods
  The test-retest reliability of MESA will be evaluated at the screening and baseline period with about one- to two-week interval among women with urgency-predominant mixed urinary incontinence.
The responsiveness of MESA questionnaire | baseline, week 12
  The responsiveness of MESA questionnaire will be evaluated before and after the treatment among women with urgency-predominant mixed urinary incontinence compared with 3-day voiding diary and ICIQ SF.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Study Chair — Guang An Men Hospital
Locations (1):
- Guang An Men Hospital, Beijing, China

REFERENCES:
- [Derived] Sun Y, Liu Y, Su T, Yuan J, Liu Z. Medical, epidemiologic, and social aspects of aging urinary incontinence questionnaire: Study protocol for the translation and validation of a Chinese language version. Medicine (Baltimore). 2019 Nov;98(44):e17719. doi: 10.1097/MD.0000000000017719. PMID 31689809